CLINICAL TRIAL: NCT01095159
Title: Comparative Study of TVTO™ X TVTS ™ for Treatment of Stress Urinary Incontinence
Brief Title: TVTO™ X TVTS ™ for Treatment of Stress Urinary Incontinence
Acronym: TVTOxTVTS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, Ana Maria Homem de Mello Bianchi, MD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNIFESP-TVTOxTVTS
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Stress Urinary Incontinence
Keywords: TVTO; TVTSecur; Mini sling; stress urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TVT-O (Active Comparator): Subjects of this group were submitted to surgical treatment of stress urinary incontinence with a transobturator sling TVT-O™ (Gynecare™, USA).
  Interventions: Device: TVT-O
- TVT-S (Active Comparator): Subjects of this group were submitted to surgical treatment of stress urinary incontinence with a transobturator mini-sling; TVT-Secur™ (Gynecare™, USA).
  Interventions: Device: TVT-S

INTERVENTIONS:
Device: TVT-O — Subjects of this group were submitted to surgical treatment of stress urinary incontinence with a transobturator sling TVT-O™ (Gynecare™, USA).
  Other Names: TVT-O™ (Gynecare™, USA).
  Arms: TVT-O
Device: TVT-S — Subjects of this group were submitted to surgical treatment of stress urinary incontinence with a transobturator mini-sling; TVT-Secur™ (Gynecare™, USA).
  Other Names: TVT-Secur™ (Gynecare™, USA).
  Arms: TVT-S

SUMMARY:
This is a prospective, comparative randomized controled trial. The general purposes of this study is to compare the efficacy and safety of TVTO™ and TVTSecur™ as surgical treatment for female urinary stress incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and urodynamic for stress urinary

Exclusion Criteria:

* Detrusor overactivity (urodynamic study)
* Urodynamic changes suggesting reduced vesical capacity
* Associated neurological diseases
* Coagulopathies
* Pregnancy
* Foreign matter sensitiveness history
* Acute urinary tract infection
* Sequel from high ionizing radiation exposure
* Use of drugs that may result in high surgical risk and/or significant postoperative complication
* Anesthetic procedure contraindication
* Vulvovaginitis: presence of vaginal secretion with infection clinically or lab supported

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2009-02; Primary Completion 2011-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Compare the efficacy of employing the Gynecare TVT Secur™ with the traditional Gynecare TVT- O™ for treating female stress urinary incontinence. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ana Maria HM BIANCHI, FELLOW, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo - Unifesp, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Carter E, Johnson EE, Still M, Al-Assaf AS, Bryant A, Aluko P, Jeffery ST, Nambiar A. Single-incision sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2023 Oct 27;10(10):CD008709. doi: 10.1002/14651858.CD008709.pub4. PMID 37888839
- [Derived] Bianchi-Ferraro AM, Jarmy-DiBella ZI, de Aquino Castro R, Bortolini MA, Sartori MG, Girao MJ. Randomized controlled trial comparing TVT-O and TVT-S for the treatment of stress urinary incontinence: 2-year results. Int Urogynecol J. 2014 Oct;25(10):1343-8. doi: 10.1007/s00192-014-2352-7. Epub 2014 Mar 19. PMID 24643378
- [Derived] Bianchi-Ferraro AM, Jarmy-Di Bella ZI, Castro Rde A, Bortolini MA, Sartori MG, Girao MJ. Single-incision sling compared with transobturator sling for treating stress urinary incontinence: a randomized controlled trial. Int Urogynecol J. 2013 Sep;24(9):1459-65. doi: 10.1007/s00192-012-1998-2. Epub 2012 Dec 4. PMID 23208003